CLINICAL TRIAL: NCT03471013
Title: Impact of Caregiver Beliefs on Adherence to Antipsychotic Medications in Patients With Schizophrenia
Acronym: CroyAid-SCZ
Status: Terminated | Type: Observational
Why Stopped: difficulty of recruitement
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-384; 2017-A02271-52 (Other: 2017-A02271-52)
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: DSM-5 Schizophrenia
Keywords: schizophrenia; beliefs; caregiver
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients and caregivers: Patients suffering from schizophrenia accompanied by their caregiver

SUMMARY:
Only one third of patients with schizophrenia are observant to their treatment knowing that the lack of adherence to treatment is one of the most important predictors of relapse.

Recent work shows that the erroneous or negative beliefs of patients with schizophrenia regarding antipsychotic treatment are associated with poor compliance.

The hypothesis is that negative beliefs about the antipsychotic treatment of caregivers of patients with schizophrenia may be associated with a higher risk of poor compliance compared to caregivers with positive beliefs about treatment.

The primary purpose is to explore the correlation between caregiver beliefs about treatment and patient compliance, taking into account the level of caregiver-patient link.

DETAILED DESCRIPTION:
Non-interventional cross-sectional exploratory study with a single visit for patients with schizophrenia and their caregivers, who agreed to participate in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* With a diagnosis of schizophrenia according to DSM-5 criteria
* Accompanied by his main caregiver, who will be able to complete the questionnaires after having signed the information form.
* Treated with one or more antipsychotics.
* Able to complete the questionnaires related to the protocol
* Having agreed to sign the information form.

Exclusion Criteria:

* Not understanding French, unable to answer questions linguistically
* Presenting an organic pathology and / or cognitive deterioration likely to hinder a good understanding of the interview
* Having already participated in the study
* presenting disorders related to the use of substances of severe intensity (such as acute intoxication, withdrawal syndrome or any state of delirium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of scizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the correlation between caregiver beliefs about treatment and patient compliance | At day 1
  The caregiver beliefs are evaluated by the Beliefs about Medicines Questionnaire, the patient compliance is evaluated by the investigator with Behaviourally Anchored Rating Scales and by the patient him-self with Morisky Medication Adherence Scale, and the level of caregiver-patient link is evaluated with Involvement Evaluation Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic SAMALIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France